CLINICAL TRIAL: NCT00393549
Title: NeuroPath Comparative Validation Study Plan
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor decision to terminate.
Sponsor: Excel-Tech Ltd. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VALP-000986
Record Dates: First submitted 2006-10-27; First posted 2006-10-30 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2007-06

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: Median Neuropathy at the wrist (MNW)
MeSH Terms: conditions — Carpal Tunnel Syndrome

INTERVENTIONS:
Device: NeuroPath

SUMMARY:
The purpose of the study is to compare the performance of the NeuroPath automated nerve conduction test with the standard of care manual test in the diagnosis of entrapment neuropathies.

ELIGIBILITY:
Symptomatic Inclusion Criteria:

* sensory symptoms (numbness and/or tingling) in at least 2 of digits 1,2,3 and 4, in at least one hand, for at least 1 month, prior to the start of the clinical study. The sensory symptoms may be intermittent or constant, but if constant, there must have been a period of time during which the symptoms were intermittent. The numbness and tingling may be accompanied by pain, but pain alone is not sufficient to meet this first inclusion criteria.
* Sensory symptoms (numbness and/or tingling) aggravated by at least 1 of the following: sleep, sustained hand or arm positioning, or repetitive actions of the hand.
* Sensory symptoms (numbness and/or tingling) mitigated by at least 1 of the following: changes in hand posture, shaking the hand, or use of a wrist splint.
* If pain is present, the wrist, hand, and finger pain is greater than elbow, shoulder, or neck pain if there is pain in any or all of those locations.

Symptomatic Exclusion Criteria:

* Sensory symptoms exclusive or predominatly in the little finger (D5) (ulnar neuropathy).
* Neck pain or shoulder pain preceded the paresthesia in the digits (cervical radiculopathy and/or brachial plexopathy).
* Numbness and/or tingling in the feet that preceded or accompanied the sensory symptoms in the hands (polyneuropathy).
* Medical history and physical examination that indicates an explanation for the sensory symptoms which is more probable than CTS. For example, digital neuropathy, median nerve pathology proximal to the carpal tunnel, ulnar neuropathy, radical neuropathy, brachial plexopathy, cervical radiculopathy, spinal cord, brainstem or brain pathology, or a polyneuropathy.
* Absence of 1st, 3rd, 4th or 5th digits
* Open wounds at the measurement sites
* Excessive sensitivity to electrical stimulation
* Median nerve injection in the past 30 days
* Prior carpal tunnel surgery
* Patients who are susceptible to radio frequency noise - such as patients with pacemakers or patients that have electrical stimulators of any sort.

Control Subject Inclusion Criteria:

* Normal neurological examination

Control Subject Exclusion Criteria:

* Absence of 1st, 3rd or 5th digits
* Open wounds at the measurement sites
* Excessive sensitivity to electrical stimulation
* Median nerve injection in the past 30 days
* Prior carpal tunnel surgery
* Reported history of CTS, polyneuropathy, diabetes,renal failure, thyroid disease or Vitamin B 12 deficiency
* Patients who are susceptible to radio frequency noise-such as patients with pacemakers or patients that have electrical stimulators of any sort.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2006-08; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Validity of the NeuroPath

SECONDARY OUTCOMES:
Accuracy of the NeuroPath

CONTACTS AND LOCATIONS:
Overall Officials: Ron Kurtz, Study Director — Excel-Tech Ltd. (XLTEK)
Locations (2):
- United States (2):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - SunCoast Neuroscience Associateion, St. Petersburg, Florida